CLINICAL TRIAL: NCT04185558
Title: Multi-Center, Prospective, Randomized, Controlled, Trial, Comparing the Safety and Efficacy of ActiGraft Pro™ to Standard of Care in Patients With Chronic Neuropathic Diabetic Foot Ulcers
Brief Title: Safety and Efficacy of ActiGraft Pro Compared to Standard of Care in DFUs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RedDress Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RD006
Record Dates: First submitted 2019-11-12; First posted 2019-12-04 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Diabetic Foot; Chronic Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- ActiGraft (Experimental): Whole blood clot (WBC) gel
  Interventions: Device: ActiGraft
- Standard of Care (Active Comparator): Alginate dressing, a non-adherent foam dressing, and an outer gauze wrap
  Interventions: Device: Standard of Care

INTERVENTIONS:
Device: ActiGraft — Whole Blood Clot (WBC) gel
  Arms: ActiGraft
Device: Standard of Care — Alginate dressing, a non-adherent foam dressing, and an outer gauze wrap
  Arms: Standard of Care

SUMMARY:
* The study is a multi-center, prospective, randomized, controlled, single blinded clinical study consisting of 150 subjects from up to 20 centers.
* The subjects are randomized to receive 1 of 2 treatments, either with ActiGraft and standard of care (SOC) or with SOC alone.
* The target ulcers are evaluated weekly by the investigator. The subject is treated once a week, to receive weekly applications of the ActiGraft + SOC or SOC until for up to 12 weeks or until the study ulcer has completely healed (i.e., 100% closure as assessed by the Investigator and blinded assessor and confirmed 2 weeks later at the healing confirmation visit (HCV). One additional visit per week is optional for both arms, for the purpose of changing only (1) the secondary dressing in the ActiGraft arm or (2) change the standard of care dressing in the control arm.
* Immediately after the study ulcer is confirmed as completely healed, subjects will enter the 12-week Follow-up Phase. During the Follow-Up phase, subjects will be evaluated twice during the first month and then monthly for two additional visits every 4 weeks until the completion of the 12-week Follow-up Phase.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥19 years of age and has type 1 or 2 diabetes
* Chronic neuropathic DFU, located distal to the malleolus (excluding ulcers between the toes but including those of the heel) and depth ≤ 5 mm with no exposed capsule, tendon or bone and no tunneling, undermining or sinus tracts (Minor tunneling and undermining will be included).
* Ulcer size between 1 cm2 and 28 cm2 (post-debridement).
* For subjects with potentially multiple eligible DFUs, the largest non-healing wound will be selected.
* Ulcer duration of ≥ 30 days. Time 0 for ulcer duration of ≥ 30 days is defined as the first day of screening (i.e., day -14). Subjects will need to meet all inclusion criteria, including lack of ulcer healing until randomization day.
* Study ulcer separated from other ulcers by at least 1 cm.
* Ulcer or affected limb free of clinical signs of infection.
* Post-debridement, ulcer free of necrotic tissue.
* Adequate circulation to the affected extremity as demonstrated by at least one of the following: (1) Transcutaneous oxygen test (TcPO2) ≥ 30 mm Hg,; (2) Ankle Brachial Index (ABI) between 0.7 and 1.2; (3)Triphasic or biphasic Doppler arterial waveforms at the ankle of affected leg; (4) Toe Brachial Index > 0.6
* HbA1c ≤ 12.0%
* Demonstrated adequate offloading regimen.
* Subject must be willing to comply with the protocol including having blood drawn to create the ActiGraft.
* Female subjects who are capable of conceiving and all males capable of insemination must use an acceptable form of contraception in order to participate in the study

Exclusion Criteria:

* Ulcer not of neuropathic diabetic foot pathophysiology (e.g., venous, vasculitic, radiation, rheumatoid, collagen vascular disease, or arterial etiology, or pressure ulcers.).
* Known or suspected ulcer malignancy of the index ulcer.
* Active Charcot of the affected foot
* Presence of underlying osteomyelitis.
* Subject with a proven sepsis established by a blood culture in the past 2 weeks, or confirmed active infection likely to interfere with trial, such as urine tract infection.
* History of alcohol or substance abuse, within the previous 2 months
* Subject has participated in another clinical trial involving a device or a systemically administered investigational study drug or treatment within 30 days of randomization visit.
* Subject is currently receiving (i.e., within the past 30 days) or scheduled to receive a medication or treatment which, in the opinion of the Investigator, is known to interfere with, or affect the rate and quality of, wound healing (e.g., systemic steroids (more than 10mg per day), immunosuppressive therapy, autoimmune disease therapy, cytostatic therapy within the past 12 months, dialysis, radiation therapy to the foot, planned vascular surgery on the study ulcer limb on the 90 days from screening, angioplasty or thrombolysis, chemotherapy).
* Subject has been treated with wound dressings that include growth factors, engineered tissues or skin substitutes (e.g., Regranex®, Dermagraft®, Apligraf®, GraftJacket®, OASIS®, Primatrix®, Matristem®, etc.) within 30 days of randomization or is scheduled to receive during the study.
* Subject has been treated with hyperbaric oxygen within 5 days of screening or is scheduled to receive during the study.
* Wound on a subject who has a life expectancy of less than 12 months.
* Subjects who are cognitively impaired and have a healthcare proxy or those who are cognitively impaired and clearly do not understand the contents of the informed consent form.
* Cannot withdraw blood in the required amount (up to 15 mL per week) technically.
* Known coagulation problems, abnormal thrombocytes level or if heparin is given intravenously. Subjects who are taking coumadin, aspirin, Plavix (clopidogrel), Eliquis or Pradaxa will not be excluded.
* Hemoglobin anemia (< 9 g/dL).
* Subject has a history of or any of the following intercurrent illnesses or conditions that would compromise the safety of the subject, or the normal wound healing process: (1) End stage renal disease; (2)Immunosuppression; (3) Severe malnutrition; (4) Liver disease; (5) Scleroderma; (6) Acquired immune deficiency disease (AIDS) or HIV positive; (7) Active connective tissue disorder; (8)Exacerbation of sickle cell anemia
* If ulcer area decreases by ≥ 30% during the initial 2-week screening (± 2 days) and standard of care phase, subject will be excluded.
* Women who are pregnant or currently breast feeding.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Incidence of complete wound closure by 12 weeks | 12 weeks
  Incidence of complete wound closure by 12 weeks using chi square (two-sided; alpha set at .05 level of significance), or Fischer exact test if one group has ≤ 5 completely closed wounds. Analysis will be adjusted using generalized linear modeling (logit function).

SECONDARY OUTCOMES:
Time to complete wound closure | 12 weeks
  Time to complete wound closure using Cox regression
Percent area reduction (PAR) | 4 weeks and 8 weeks
  Percent area reduction (PAR) at 4 and 8 weeks.
Nature, frequency, and severity of adverse events in the intent to treat population | 12 weeks
  Nature, frequency, and severity (by CTCAE5) of adverse events
Number of patients showing a consistence wound closure post healing determination | 24 weeks

CONTACTS AND LOCATIONS:
Locations (16):
- United States (12):
  - Institute for Advanced Wound Care, Montgomery, Alabama
  - New Hope Podiatry Group Inc, Los Angeles, California
  - Greater Los Angeles VA, Los Angeles, California
  - Center for Clinical Research Inc, San Francisco, California
  - Olive View UCLA Education & Research Institute, Sylmar, California
  - Eric J Lullove DPM PA, Coconut Creek, Florida
  - Future Health Research Clinic, Miami, Florida
  - Barry University Clinical Research, North Miami Beach, Florida
  - Pacific Vascular Institute, Hilo, Hawaii
  - Boston Medical Center, Boston, Massachusetts
  - Wahab Consulting and Research LLC, Las Vegas, Nevada
  - Temple University, Philadelphia, Pennsylvania
- South Africa (3):
  - Wound Care South Africa, Germiston
  - Haute Care, Lyttelton
  - Eloquent Health & Wellness, Tyger Valley
- Acinadem Altunizade, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No